CLINICAL TRIAL: NCT04120584
Title: Clinical Evaluation of Safety and Efficacy of Radio Frequency (Forma Eye) Treatment for Dry Eye Disease Due to Meibomian Gland Dysfunction
Brief Title: Radio Frequency (Forma Eye) Treatment for Dry Eye Disease Due to Meibomian Gland Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO609175A
Record Dates: First submitted 2019-10-04; First posted 2019-10-09 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2024-06

CONDITIONS: Improvement of Dry Eye Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Forma Eye treatment (Experimental)
  Interventions: Device: Forma Eye Applicator

INTERVENTIONS:
Device: Forma Eye Applicator — Eligible subjects will receive up to 3 treatments (2-3 weeks interval) with the Forma Eye Applicator according to the study protocol.
  The subject will return for 3 follow up visits: four weeks (4wk FU), 12 weeks (12wk FU), twenty-four weeks (24wk FU) after the last treatment.

SUMMARY:
The aim of the study is to evaluate the safety and efficacy of radiofrequency treatment for dry eye disease due to meibomian gland dysfunction

ELIGIBILITY:
Inclusion Criteria:

1. Adult females and males between the ages of 18 -75, seeking treatments for Dry Eye Disease Due to Meibomian Gland Dysfunction
2. Tear breakup time (TBUT) ≤10 s;
3. Evidence of meibomian gland (MG) obstruction, based on total MGS of ≤12 in lower eyelids for each eye as assessed by a clinician not involved in the study procedure
4. Subjective symptom score (using the Standard Patient Evaluation of Eye Dryness [SPEED] questionnaire) ≥10;
5. At least one meibomian gland opening with a visible plugging over the eyelid margin
6. No ocular pathology requiring treatment other than eye lubricant and conventional eyelid hygiene within the last month and during the study
7. The subjects should understand the information provided about the investigative nature of the treatment, possible benefits, and side effects, and sign the Informed Consent Form
8. The subjects should be willing to comply with the study procedure and schedule, including follow up visits.
9. Agreement/ability to abstain from dry eye/MGD medications or any device treatments for the time between the treatment visit and the final study visit. Ocular lubricants are allowed if no changes are made during the study.

Exclusion Criteria:

1. Evidence of co-existing ocular conditions potentially posing an increased risk of procedure-related injury, (e.g., active ocular infection or inflammation in either eye)
2. History of ocular trauma or surgery including intraocular, oculoplastic, corneal or refractive surgery within 1 year
3. Ocular surface abnormality potentially compromising corneal integrity in either eye; eyelid abnormalities affecting lid function in either eye
4. Systemic disease conditions that cause dry eye (e.g., Stevens-Johnson syndrome, vitamin A deficiency, rheumatoid arthritis, Wegener's granulomatosis, sarcoidosis, leukemia, Riley-Day syndrome, systemic lupus erythematosus, Sjogren's syndrome)
5. Unwillingness to abstain from systemic medications known to cause dryness for the study duration.
6. Individuals who have either changed the dosing of systemic or non-dry eye/MGD ophthalmic medication within the past 30 days prior to screening
7. Internal defibrillator, a pacemaker or any other implanted electrical device anywhere in the body
8. Permanent metal implant in the treatment area
9. Any surgery in the treatment area in the last 3 months
10. Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles
11. Pregnancy and nursing or females of childbearing potential and not utilizing adequate birth control measures
12. Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications
13. Patients with a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
14. Poorly controlled endocrine disorders, such as diabetes, thyroid dysfunction, polycystic ovary, and hormonal virilization
15. Any active condition in the treatment area, such as but not limited to open sores, psoriasis, eczema, vitiligo, herpes, and rash.
16. History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin
17. Severe concurrent conditions, such as cardiac disorders, sensory disturbances.
18. Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
19. Participation in another study within 30 days prior to screening.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Paul, MD, Principal Investigator — 4316 James Casey St Building F Suite 201, Austin, TX 78745, United States; Sandy Zhang-Nunes, MD, Principal Investigator — Oculofacial Plastic Surgery Director USC Roski Eye Institue USC Keck School of Medicine
Locations (3):
- United States (3):
  - Centennial Eye Associates, Aurora, Colorado
  - Excellent Vision, Portsmouth, New Hampshire
  - Sean Paul, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Forma Eye treatment: Forma Eye Applicator: Eligible subjects will receive up to 3 treatments in both eyes (2-3 weeks interval) with the Forma Eye Applicator according to the study protocol.
  The subject will return for 3 follow up visits: four weeks (4wk FU), 12 weeks (12wk FU), twenty-four weeks (24wk FU) after the last treatment.
Period: Overall Study
Arm/Group | Forma Eye treatment
Started | 47
Completed | 35
Not Completed | 12

BASELINE CHARACTERISTICS:
Groups:
- Forma-Eye treatment: Eligible subjects will receive up to 3 treatments in both eyes(2-3 weeks interval) with the Forma Eye Applicator according to the study protocol.
Arm/Group | Forma-Eye treatment
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 47.79 [23 to 75]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 47 included 35 complete the study
  Participants
    Female | 27
    Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Standardized Patient Evaluation of Eye Dryness (SPEED) [Mean (Standard Deviation); unit: score on scale] — Standard Patient Evaluation of Eye Dryness Questionnaire (SPEED) The SPEED questionnaire was designed to quickly track the progression of dry eye symptoms over time. This questionnaire gives a score from 0 to 28 that is the result of 8 items that assess frequency and severity of symptoms.0-4: mild, 5-7: moderate, 8+: severe
  score on scale | 15.647 (4.7)
Meibomian Gland Score (MGS), as Assessed by a Masked Rater [Mean (Standard Deviation); unit: score on a scale]
  Right Eye | 6 (4.17)
  Left Eye | 5.32 (3.13)
Tear Break-Up Time [Mean (Standard Deviation); unit: score on a scale]
  Right eye | 2.77 (1.56)
  Left eye | 2.9 (2.06)
Ocular Surface Disease Index (OSDI) [Mean (Standard Deviation); unit: score on scale] | 34.5 (18.6)
Corneal Surface fluorescent staining using NEI (National Eye Institute) grading [Mean (Standard Deviation); unit: score on a scale]
  Right eye | 2.7 (1.15)
  Left eye | 2.85 (1.51)

OUTCOME MEASURES:

1. Primary Outcome: Standardized Patient Evaluation of Eye Dryness (SPEED)
Description: Change dry eye symptoms evaluated by Standardized Patient Evaluation of Eye Dryness (SPEED) This questionnaire gives a score from 0 to 28. Lower score indicates better outcome. 0-4: mild, 5-7: moderate, 8+: severe Scale range: 0 (minimum; no symptoms) to 28 (maximum; most severe symptoms). Interpretation: Lower scores indicate better outcomes. Symptom severity can be categorized as: 0-4 = mild, 5-7 = moderate, 8-28 = severe.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Forma Eye treatment
Number analyzed (Participants) | 35
score on a scale | 9.6 (5.79)
Statistical Analysis 1: Comparison: Forma Eye treatment; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = 9.62

2. Primary Outcome: Meibomian Gland Score (MGS), as Assessed by a Masked Rater
Description: The Meibomian Gland Score (MGS) is a standardized clinical tool used to assess the functional quality of the meibomian glands, which are responsible for secreting the oily layer of the tear film. Dysfunction in these glands is a common cause of dry eye disease and evaporative dry eye. The scoring typically involves gentle expression of the meibomian glands, usually from a designated number of glands (commonly 15, e.g., 5 each from the nasal, central, and temporal parts of the lower eyelid). Each gland is evaluated based on the quality of the secretion it produces.
  Scoring Criteria per Gland:
  Each gland is scored on a 0-3 scale:
  0 = No secretion
  1. = Inspissated/toothpaste-like secretion
  2. = Cloudy secretion
  3. = Clear, healthy oil
  If 15 glands are assessed, the maximum total score is 45 (15 glands × 3 points per gland).
  A higher total MGS reflects better meibomian gland function and healthier tear film, indicating a more favorable condition.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Forma Eye treatment
Number analyzed (Participants) | 35
score on a scale
  Right eye | 21.8 (11.26)
  Left Eye | 23.9 (12.84)
Statistical Analysis 1: Comparison: Forma Eye treatment; Test type: Superiority; p < 0.001, ANOVA

3. Primary Outcome: Tear Break-Up Time
Description: Tear Break-Up Time (TBUT) Changes in dry eye symptoms such as ocular fatigue or dryness will be assessed by TBUT. The measurement is reported in seconds.
  * Scale range: 0 seconds (minimum) to >10 seconds (maximum normal value considered).
  * Interpretation: >10 seconds = normal, 5-10 seconds = marginal, <5 seconds = low.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Forma Eye treatment
Number analyzed (Participants) | 35
seconds
  Right eye | 7.1 (3.50)
  Left eye | 7.055 (2.76)

4. Primary Outcome: Ocular Surface Disease Index (OSDI)
Description: Ocular Surface Disease Index (OSDI) This 12-item questionnaire assesses dry eye symptoms and their effects. Scale range: 0 (minimum) to 100 (maximum). Interpretation: Lower scores indicate better outcomes.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Forma Eye treatment
Number analyzed (Participants) | 35
score on a scale | 23.5 (18.59)

5. Primary Outcome: Corneal Surface Fluorescent Staining Using NEI (National Eye Institute) Grading
Description: Change in measurements using ocular surface fluorescent staining. The NEI scale divides the corneal and conjunctival surfaces to grade fluorescein uptake. Each of 5 areas per cornea is graded 0-3. The NEI scale for grading fluorescein staining divides the corneal and conjunctival surfaces to help measure fluorescein uptake. A standardized grading system of 0 to 3 is used for each of the five areas on each cornea.
  Scale range: 0 (minimum; no staining) to 15 (maximum). Interpretation: Lower scores indicate better outcomes.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Forma Eye treatment
Number analyzed (Participants) | 35
score on a scale
  Right eye | 0.18 (0.77)
  Left eye | 0.8 (0.19)

6. Secondary Outcome: Subject's Assessment of Improvement
Description: Subject assessment of improvement based on 0 - 4-point Likert scale. Improvement assessment will be performed independently by the subject himself on the following 0-4 points Likert scale questionnaire (Global Aesthetic Improvement Scale):
  4 = Significantly marked improvement; 3 = Marked improvement; 2 = Moderate improvement; 1 = Slight improvement; 0 = No difference Scale range: 0 (no difference) to 4 (significant marked improvement).
Time Frame: 6 months
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Forma Eye treatment
Number analyzed (Participants) | 35
score on a scale | 1.71 (1.48)

7. Secondary Outcome: Subject Assessment of Satisfaction
Description: Subject assessment of satisfaction will be filled-out by subjects only using 5-points Likert scale:
  +2 = Very satisfied; +1 = Satisfied; 0 = Indifferent; -1 = Disappointed; -2 = Very disappointed.
  Scale range: -2 (very disappointed) to +2 (very satisfied). Interpretation: Higher scores indicate better outcomes.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Forma Eye treatment
Number analyzed (Participants) | 35
score on a scale | 1 (0.87)

8. Secondary Outcome: Safety Assessment
Description: Discomfort assessment during the treatment using NSR scale. At each treatment the subject will be asked to fill assessments for the pain/discomfort during the procedure. The subject will be asked to rate the severity from 0 to 10, with 0 equaling no symptoms and 10 equaling the worst possible symptoms. A number is obtained by measuring up to the point the subject has indicated.
  Scale range: 0 (no pain) to 10 (worst possible pain).
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Forma Eye treatment
Number analyzed (Participants) | 35
units on a scale | 1.6 (1.9)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Forma Eye treatment
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 2/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Forma Eye treatment (N=47)
conjuctivitis (Eye disorders) | 1 (1)
swollen lids (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT04120584/Prot_SAP_000.pdf